CLINICAL TRIAL: NCT06399653
Title: Non-invasive Vagal Nerve Stimulation as Novel Treatment to Improve Functional Outcomes in Veterans With Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N4777-M
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; neuromodulation; neuroimaging; withdrawal; anxiety; autonomic nervous system
MeSH Terms: conditions — Alcoholism; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either active or placebo stimulation, and will receive identical instructions on use of the device. Participants will remain in the same condition assigned at baseline and will be instructed to self-administer nVNS/sham at home for 7 days (2 mins bilaterally, 2x per day) and return for a follow-up visit. Stimulation will be administered by the examiner during a functional MRI scan during the baseline and the follow-up visit.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Devices will be masked to ensure both the research team involved in data collection and participants are blinded (double-blind study design). An unblinded member of the research team, not involved in data collection and subject contact, will assign randomization, provide device identification number, and keep the key linking condition to identification numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active cervical transcutaneous vagus nerve stimulation (Active Comparator): Participants will be assigned to active transcutaneous vagus nerve stimulation, received once during each of the study visits and self-administered twice a day for a week.
  Interventions: Device: Cervical transcutaneous vagus nerve stimulation (active comparator)
- Sham cervical transcutaneous vagus nerve stimulation (Placebo Comparator): Participants will be assigned to sham transcutaneous vagus nerve stimulation, received once during each of the study visits and self-administered twice a day for a week.
  Interventions: Device: Cervical transcutaneous vagus nerve stimulation (sham comparator)

INTERVENTIONS:
Device: Cervical transcutaneous vagus nerve stimulation (active comparator) — Active nVNS produces low-voltage electrical signal that generates sensations on the skin on upper anterior cervical area (overlying carotid artery) and that stimulates the vagus nerve.
  Other Names: gammaCore
  Arms: Active cervical transcutaneous vagus nerve stimulation
Device: Cervical transcutaneous vagus nerve stimulation (sham comparator) — Sham nVNS devices look identical to active devices and participants will undergo identical training for self-administration on upper anterior cervical area (overlying carotid artery). Sham devices do not stimulate the vagus nerve.
  Other Names: sham
  Arms: Sham cervical transcutaneous vagus nerve stimulation

SUMMARY:
Alcohol use disorder (AUD) is a major health concern amongst Veterans as it causes functional impairments and decreased quality of life. Current AUD treatments show limited effectiveness in reducing withdrawal-related psychological and physical distress, which drives the urge to drink to relieve these symptoms. The investigators propose the vagus nerve, which is the primary nerve of the "rest and digest" branch of the autonomic nervous system via its bidirectional connections between the brain and the body, as a novel treatment target for AUD. The goal of this study is to assess treatment efficacy and mechanism of action. Noninvasive neuromodulation technologies offer the possibility for innovative, low risk treatments to support the rehabilitation and community reintegration of Veterans with AUD.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a serious mental health disorder that affects more than 40% of US military Veterans, presenting a major burden to this population and to the VA Healthcare System. Relapse rates of AUD are extremely high; over half of Veterans who complete treatment, relapse within 6 months, highlighting the need for improved treatments or different treatment targets. Long-term excessive drinking results in homeostatic dysregulation due to changes in the central and autonomic nervous system, which manifests in psychological and physical distress during abstinence and results in the urge to drink to relieve these symptoms. These symptoms, which can be equated to withdrawal, lead to continued harmful drinking and relapse, and are associated with significant functional impairment and reduced quality of life.

Current AUD treatments do not effectively mitigate this homeostatic dysregulation and have risks and side effects as well as other limitations. The investigators propose the vagus nerve, which is the main nerve of the parasympathetic branch of the autonomic nervous system and plays an important role in maintaining and restoring physiological homeostasis, as a novel treatment target for AUD. Noninvasive stimulation of the vagus nerve (nVNS) has been shown to alleviate anxiety, depression, and pain. The investigators hypothesize that nVNS can restore homeostasis and reduce withdrawal-related distress and craving, and consequently improve functional outcomes and quality of life in Veterans with AUD.

The goal of this study is to assess treatment efficacy and mechanism of action. The proposed study will include 80 Veterans with current AUD, who will be randomized to receive nVNS or sham stimulation prior to performing a well-validated heat pain task designed to assess neural and physiological correlates of distress. Subjects will then self-administer nVNS/sham at home twice a day for 7 days and return for a follow-up visit, during which all study components will be repeated. Behavioral assessments of psychological and physiological distress, craving, and functional outcomes will be administered at baseline and post-treatment, as well as at a 1-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans between 21 and 65 years, any race or ethnicity.
2. Meet current DSM-5 diagnosis of moderate or severe AUD (Structured Clinical Interview for DMS-5 (SCID) interview) with at least one functional disability due to alcohol use, current alcohol craving, and current heavy drinking (>= 5 drinks (men) / >= 4 drinks (women) on the same occasion, on 5 or more days in the past month) as defined by the Substance Abuse and Mental Health Services Administration (SAMHSA), and mild to moderate withdrawal symptoms during abstinence.
3. Able to forgo consumption of alcohol for 12-24 hours without any serious discomfort or complications.
4. Capable of complying with study schedule, procedures, and speaks English.
5. Able to provide voluntary written informed consent prior to initiation of visit 1.
6. Able and willing to self-administer nVNS/sham stimulation as instructed for the duration of the study, and willing to commit to the return visit at the end of the study.

Exclusion Criteria:

1. Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-Ar) score >10 on the day of the scan (symptoms judged to be due to co-existing anxiety or headache disorders will not be counted toward the total).
2. Recent history past 6 months) of severe complications due to alcohol withdrawal (alcohol withdrawal seizures, hallucinations/illusions, delirium tremens).
3. Currently or recently (within last 90 days) enrolled in abstinence-based treatment program.
4. Evidence of a maladaptive pattern of substance use or abuse other than alcohol one month prior to screening visit.
5. Uncontrolled severe psychiatric disorder with psychotic symptoms or cognitive impairment. We will not exclude for PTSD.
6. At risk for suicide requiring urgent higher-level care or homicide (based on the Columbia-Suicide Severity Rating Scale and follow-up clinical interview).
7. History of neurological disorder that might be associated with cognitive dysfunction.
8. History of head trauma involving loss of consciousness >24 hours
9. Clinically significant uncontrolled/unstable medical illness or clinically significant surgery within 1 month of the screening visit.
10. MRI-related exclusion criteria: cardiac pacemaker, metal fragments in eyes/skin/body, aortic/aneurysm clips, heart-valve replacement, copper intrauterine device, shunt (ventricular or spinal), neuro/bio-stimulators, (for females) pregnant or nursing. Any implants will be reviewed for safety.
11. Vagus nerve stimulation related criteria: active implantable medical device, metallic device implanted at or near the neck, carotid atherosclerosis (narrowing of arteries), cervical vagotomy, clinically significant hypertension, hypotension, bradycardia, or tachycardia, cardiac disease and atherosclerotic cardiovascular disease (severe carotid artery disease (e.g., history of transient ischemic attack (TIA) or stroke), congestive heart failure, severe coronary artery disease or recent myocardial infarction (within 5 years)).
12. Pharmacotherapy for AUD: >= 2 weeks stability is required to ensure a steady state of medication effects prior to nVNS administration.
13. Currently taking opioids or benzodiazepines.
14. In case it is determined by the investigator during the course of the study, that a subject needs a higher level or care, study participation will be discontinued, and the subject will be excluded from the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The HAM-A is a 14-item scale that assesses the presence and severity of psychological distress and negative emotional states. Completion takes 10 minutes. This instrument is widely used in clinical trials and alcohol studies and is sensitive to both nVNS and AUD treatment. Items are rated on a scale ranging from 0 (not present) to 4 (very severe).
Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) is a short form (5 min.) to assess symptoms of acute alcohol withdrawal and physical discomfort. The CIWA-Ar includes 8 items, 7 of which are rated from 1 to 7 (higher score indicating higher severity) and 1 of which is rated from 0 to 4 (higher score indication less orientation to place/or person)
Alcohol Urge Questionnaire (AUQ) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The Alcohol Urge Questionnaire (AUQ) is 8-item scale that measures cognitive preoccupation with alcohol on a 7-point rating scale ranging from "strongly disagree" to "strongly agree". Two items are reverse scored. Higher scores reflect greater craving.
WHO Quality of Life assessment (WHOQOL-BREF) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The WHOQOL-BREF assesses quality of life across four domains (physical health, psychological, social relationships, and environment) with a total of 26 questions. The WHOQOL-BREF is a widely used instrument with strong psychometric properties.

SECONDARY OUTCOMES:
Neural response to heat pain fMRI task | Baseline to week 1 of 2x daily intervention
  During this task, participants receive brief thermal stimuli (experienced temperature ranging from warm to hot) applied to the leg via a thermode. Neural activation will be measured using percent signal change with higher scores indicating greater activation.

OTHER OUTCOMES:
Physiological response to heat pain fMRI task | Baseline to week 1 of 2x daily intervention
  During this task, participants receive brief thermal stimuli (experienced temperature ranging from warm to hot) applied to the leg via a thermode. Autonomic response to will be indexed by galvanic skin response and heart rate variability.
The Drinker Inventory of Consequences (DrInC) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The DrInC assesses adverse alcohol-related consequences; the first administration establishes consequences in the past 30 days, and second administration assesses post-treatment problems.
Substance Use Recovery Evaluator (SURE) | Baseline to week 1 and 1 month post baseline of 2x daily intervention
  The Substance Use Recovery Evaluator (SURE) assesses the following domains of AUD-related functional outcomes: self-care (mental and physical health), relationships, material resources (stability of housing and occupational resources), and outlook of life. The SURE has been developed for use in substance use disorder populations. The SURE is comprised of 21 items, rated on a 3-point scale, but scored using a 3-point scale. Scores range from 21-63.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Klaming, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No